CLINICAL TRIAL: NCT05815706
Title: The Effect of the Supplemental Nursing System-Based Feeding on Time to Transition to Exclusive Breastfeeding, Sucking Success, and Discharge Time: A Randomized Controlled Trial on Preterm Infants
Brief Title: The Effect of the SNS-Based Feeding on Transition to Exclusive Breastfeeding in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-1/20
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Breastfeeding; Preterm Infant; Sucking Behavior
MeSH Terms: conditions — Breast Feeding; Premature Birth; Sucking Behavior

STUDY DESIGN:
Intervention Model Description: Participants were randomized into the experimental and control groups using a block randomization method. Research shows that gestational age and sucking experience affect the sucking behavior of preterm infants (Kaya and Aytekin, 2017; Yildiz and Arikan, 2012). Therefore, gestational age (30-32 and 33-34 weeks), gender (girls and boys), and LATCH scores (0-2, 3-6, and 7-10 points) were used for block randomization. The blocks were repeated three times in each group. Thirty-six participants were assigned to each group. A 2X2X3X3 blocked randomization list was developed using an online randomization tool (Sealed Envelope Ltd, 2018).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group participants were breastfed for ten minutes (five minutes for each breast) every day from the day they started oral feeding until they switched to exclusive breastfeeding. The nurse placed the warmed breast milk or formula in SNS. She then fixed it to the mother's nipples. Each experimental group participant sucked on the two breasts for 15 minutes. Breastfeeding (ten minutes), resting and SNS preparation (five minutes), and SNS feeding (15 minutes) were limited to a total of 30 minutes in light of earlier research.
  Interventions: Device: MEDELA Supplemental nursing system
- Control (No Intervention): Preterm infants were fed according to the clinical feeding protocol. They were not SNS-fed.

INTERVENTIONS:
Device: MEDELA Supplemental nursing system — The experimental group participants were fed based on the MEDELA Supplemental Nursing System, which consists of a syringe/container and a feeding catheter. One end of the feeding probe is in the syringe/container, while the other is fixed to the mother's nipple through a plaster. MEDELA SNS is a sterile product with an adjustable breast milk flow system and neck strap. It is bisphenol A (BPA) free. All its parts are in direct contact with breast milk. This system allows the baby to both suck and feed (MEDELA Supplemental Nursing System, 2018).
  Arms: Experimental

SUMMARY:
This study investigated the effect of the Supplemental Nursing System (SNS)-based feeding on the time to transition to exclusive breastfeeding, sucking success, and the time to discharge in preterm infants

DETAILED DESCRIPTION:
Nutrition is a critical problem in preterm infants. They should initially be enterally fed because they have poor sucking-swallowing-breathing coordination. Once a preterm infant develops that coordination, enteral feeding should be discontinued immediately. Then, the preterm should switch to oral feeding (breastmilk). However, preterm infants are not good at sucking because they get tired too quickly, have poor sucking skills, and lack enough experience. Therefore, we must use alternative supplemental feeding methods (bottle, spoon, dropper, cup, breastfeeding support system, and finger feeding) until preterm infants mature enough to meet their daily nutritional needs by breastfeeding alone (exclusive breastfeeding).

The Supplemental Nursing System (SNS) is an alternative supplemental feeding method that supports the development of sucking skills while providing the preterm infant's nutritional needs. This study investigated the effect of the Supplemental Nursing System (SNS)-based feeding on the time to transition to exclusive breastfeeding, sucking success, and the time to discharge in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* being between the gestational ages of 30 to 34 weeks
* having a birthweight of ≥1000 g
* having an APGAR score of >6
* having stabilized for 48 hours after receiving mechanical ventilator or continuous positive air pressure or both
* being exclusively gavage-fed with breast and/or formula and ready to switch to oral feeding
* being willing to breastfeed

Exclusion Criteria:

* having a congenital malformation that may cause asphyxia and affect breathing
* having an intraventricular hemorrhage, intracranial hemorrhage, or periventricular leukomalacia
* having intestinal anomalies or hyperbilirubinemia requiring exchange transfusion
* having respiratory distress syndrome, bronchopulmonary dysplasia, or other chronic lung diseases.

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The time to transition to oral feeding (hours) | up to three weeks
  It was measured when the preterm infant swiched from gavage feeding to oral feeding.
Time to discharge (hours) | up to 2 months
  It was measured at discharge
The sucking success (First measurement) | at the beginning of the study, up to three weeks
  The sucking success was assessed using the LATCH Breastfeeding Assessment Tool. The tool was developed by Jensen et al. (1994) and adapted to Turkish by Yenal and Okumus (2003). It consists of five evaluation criteria: L (Latch on breast), how well the infant latches onto the breast; A (Audible swallowing), the amount of audible swallowing noted; T (Type of nipple), the mother's nipple type; C (Comfort, breast/nipple), the mother's level of comfort in relation to the nipple; and H (Hold/Help), the amount of help the mother needs to hold her infant to the breast. Each item is rated on a scale of 0 to 2. The total score ranges from 0 to 10, with high scores indicating successful sucking.
The sucking success (Second measurement) | 48 hours after the second measurement of sucking success
  The sucking success was assessed using the LATCH Breastfeeding Assessment Tool. The tool was developed by Jensen et al. (1994) and adapted to Turkish by Yenal and Okumus (2003). It consists of five evaluation criteria: L (Latch on breast), how well the infant latches onto the breast; A (Audible swallowing), the amount of audible swallowing noted; T (Type of nipple), the mother's nipple type; C (Comfort, breast/nipple), the mother's level of comfort in relation to the nipple; and H (Hold/Help), the amount of help the mother needs to hold her infant to the breast. Each item is rated on a scale of 0 to 2. The total score ranges from 0 to 10, with high scores indicating successful sucking.
The sucking success (Last measurement) | through study completion, an average of 2 months
  The sucking success was assessed using the LATCH Breastfeeding Assessment Tool. The tool was developed by Jensen et al. (1994) and adapted to Turkish by Yenal and Okumus (2003). It consists of five evaluation criteria: L (Latch on breast), how well the infant latches onto the breast; A (Audible swallowing), the amount of audible swallowing noted; T (Type of nipple), the mother's nipple type; C (Comfort, breast/nipple), the mother's level of comfort in relation to the nipple; and H (Hold/Help), the amount of help the mother needs to hold her infant to the breast. Each item is rated on a scale of 0 to 2. The total score ranges from 0 to 10, with high scores indicating successful sucking.
The time to transition to exclusive breastfeeding (hours) | up to two weeks
  It was measured when the preterm infant transitioned to exclusive breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Result] Kaya V, Aytekin A. Effects of pacifier use on transition to full breastfeeding and sucking skills in preterm infants: a randomised controlled trial. J Clin Nurs. 2017 Jul;26(13-14):2055-2063. doi: 10.1111/jocn.13617. Epub 2017 Mar 21. PMID 27754572
- [Result] Penny F, Judge M, Brownell E, McGrath JM. What Is the Evidence for Use of a Supplemental Feeding Tube Device as an Alternative Supplemental Feeding Method for Breastfed Infants? Adv Neonatal Care. 2018 Feb;18(1):31-37. doi: 10.1097/ANC.0000000000000446. PMID 29373347
- [Result] Penny F, Judge M, Brownell EA, McGrath JM. International Board Certified Lactation Consultants' Practices Regarding Supplemental Feeding Methods for Breastfed Infants. J Hum Lact. 2019 Nov;35(4):683-694. doi: 10.1177/0890334419835744. Epub 2019 Apr 19. PMID 31002761
- [Result] Celik F, Sen S, Karayagiz Muslu G. Effects of Oral Stimulation and Supplemental Nursing System on the Transition Time to Full Breast of Mother and Sucking Success in Preterm Infants: A Randomized Controlled Trial. Clin Nurs Res. 2022 Jun;31(5):891-900. doi: 10.1177/10547738211058312. Epub 2021 Nov 16. PMID 34784787
- [Result] Calikusu Incekar M, Caglar S, Kaya Narter F, Tercan Tarakci E, Ozpinar E, Demirci Ecevit E. An alternative supplemental feeding method for preterm infants: the supplemental feeding tube device. Turk J Med Sci. 2021 Aug 30;51(4):2087-2094. doi: 10.3906/sag-2009-323. PMID 33992038